CLINICAL TRIAL: NCT02878226
Title: Uterine Rupture: Prevalence and Feto-maternal Outcomes in Assiut Women Health Hospital
Brief Title: Outcomes of Uterine Rupture
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: UR
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Maternal Mortality
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: repair of rupture

SUMMARY:
Uterine rupture (UR) is a serious, life-threatening obstetric complication. UR is associated with an increased risk of maternal and perinatal morbidity and mortality, particularly in developing countries compared to developed countries. UR occurs mainly as a consequence of poorly managed labour

ELIGIBILITY:
Inclusion Criteria:

* women with ruptured uterus
* accept to share in the study

Exclusion Criteria:

* women refuse to participate

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients presented with clinical symptoms and signs of rupture uterus, whatever the duration of pregnancy, and the diagnosis proved on surgical exploration to be a case of rupture uterus
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
number of women undergoes repair | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided